CLINICAL TRIAL: NCT02119143
Title: Influence of Micronutrient Supplementation on Duty Days Lost Due to Flu/Common Cold, Immune System, Oxidative Stress and Wellbeing in a Cohort of Middle Management Employees
Brief Title: Micronutrient Supplementation and Incidence of Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Beat (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Principal Investigator, Green Beat
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 26-151 ex 13/14
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Immune System Diseases
Keywords: common cold, immunity, oxidative stress
MeSH Terms: conditions — Immune System Diseases; Common Cold | interventions — Minerals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamines and minerals (Active Comparator): 41 middel aged subjects receive vitamin and mineral supplementation
  Interventions: Dietary Supplement: vitamines and minerals
- cellulose (Placebo Comparator): 41 middle aged subjects get the placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: vitamines and minerals — given for 24 weeks, after 4 week wash out of all supplements and dietetic products
  Arms: Vitamines and minerals
Dietary Supplement: placebo — given for 24 weeks, after 4 weeks wash out of all supplements and dietetic products
  Arms: cellulose

SUMMARY:
This study investigates the effects of a dietary supplement - a cocktail of vitamins and minerals - on the incidence of common cold in a cohort of middle management employees.The primary outcome is defined as the number of duty days lost due to common cold/flu. Further, immune parameters and markers of redox biology/oxidative stress will be determined. The wellbeing in the cohort will be evaluated via questionnaires.

DETAILED DESCRIPTION:
randomized, double-blinded, placebo controlled trial 82 Subjects, men and women, 25 - 50 yrs, non-smokers, employees of middle management, 24 weeks of supplementation/placebo, 4 wk wash-out of all supplements and dietetic products, undersupply of fruit, vegetables (< 4 portions/day) and whole grain food (< 5x/wk)

ELIGIBILITY:
Inclusion Criteria:

* pre or peri-menopausal
* non-smokers
* sedentary or moderately trained
* BMI: >20 and < 35kg/m2
* undersupply of fruits, vegetables and whole grain food, fibres
* contraceptives
* wash-out

Exclusion Criteria:

* post-menopausal
* smokers
* trained people
* BMI out of inclusion range
* adequate intake of vegetables, fruits and whole grain food, fibres
* no adherence to wash-out

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-04; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Incidence of common cold | 24 weeks
  vitamins and minerals might influence the incidence of common cold in middle aged management employees

SECONDARY OUTCOMES:
change in immune markers | 24 weeks
  cytokine levels and expression of cytokine receptors in leucocytes may change over time due to micronutrient intervention

OTHER OUTCOMES:
change in redox biology | 24 weeks
  micronutrients may influence redox biology of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, Prof, Principal Investigator — Green Beat and Medical University of Graz
Locations (1):
- Institute of Pathophysiology and Immunology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No